CLINICAL TRIAL: NCT02485925
Title: The Effectiveness and Safety in the Treatment of Circumferential Pulmonary Vein Isolation (CPVI) for Symptomatic Paroxysmal Atrial Fibrillation With THERMOCOOL® SMARTTOUCH™ Catheter in China, A Multi-center Clinical Registry Study
Brief Title: SMART China, A Multi-center Clinical Registry Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BW-201501
Record Dates: First submitted 2015-06-25; First posted 2015-06-30 (Estimated); Results first posted 2018-07-31 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation
Keywords: Interventional; Radiofrequency ablation; Paroxysmal Atrial Fibrillation; Catheter ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment group (Experimental): THERMOCOOL® SMARTTOUCH™
  Interventions: Device: THERMOCOOL® SMARTTOUCH™

INTERVENTIONS:
Device: THERMOCOOL® SMARTTOUCH™ — Pulmonary vein isolation by RF ablation treatment with the THERMOCOOL® SMARTTOUCH™ contact force sensing catheters (study device)
  Other Names: Pulmonary vein isolation

SUMMARY:
This is a prospective effectiveness and safety assessment of the study device during radiofrequency (RF) ablation treatment of patients with drug refractory symptomatic atrial fibrillation.

DETAILED DESCRIPTION:
The purpose of this study is to assess the effectiveness and safety of the THERMOCOOL® SMARTTOUCH™ catheter in the treatment of drug refractory symptomatic paroxysmal atrial fibrillation (PAF) undergoing CPVI.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Failure of at least one antiarrhythmic drug (AAD) for AF (class I or III, or AV nodal blocking agents such as beta blockers and calcium channel blockers) as evidenced by recurrent symptomatic AF, or intolerance to the AAD
3. Patients with paroxysmal AF eligible for catheter ablation
4. Patients with symptomatic PAF who have had at least one documented AF episode in the twelve (12) months prior to enrollment. Documentation may include but is not limited to electrocardiogram (ECG), Holter monitor (HM) or transtelephonic monitor (TTM)
5. Able and willing to comply with all pre-, post- and follow-up testing and requirements
6. Be able to sign IRB/EC-approved informed consent form

Exclusion Criteria:

1. AF secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause
2. Previous surgical or catheter ablation for AF
3. Any PCI, cardiac surgery, or valvular cardiac surgical or percutaneous procedure (e.g., ventriculotomy, atriotomy, and valve repart or replacement and presence of a prosthetic valve) within the past 2 months.
4. Any carotid stenting or endarterectomy.
5. Coronary artery bypass graft (CABG) procedure within the last 180 days (6 months)
6. AF episodes lasting longer than 7 days or terminated via cardioversion
7. Documented left atrial thrombus on imaging
8. Uncontrolled heart Failure or New York Heart Association (NYHA) class III or IV
9. Myocardial Infarction within the previous 60 days (2 months)
10. Documented thromboembolic event (including TIA) within the past 12 months
11. Rheumatic heart disease
12. Awaiting cardiac transplantation or other cardiac surgery within the next 365 days (12 months)
13. Significant pulmonary disease, (e.g., restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease) or any other disease or malfunction of the lungs or respiratory system that produces chronic symptoms.
14. Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment in this study
15. Active illness or active systemic infection or sepsis
16. Diagnosed atrial myxoma
17. Unstable angina within the past 60 days (2 months)
18. History of blood clotting or bleeding abnormalities
19. Life expectancy less than 365 days (12 months)
20. Hypertrophic obstructive cardiomyopathy
21. Presence of implanted ICD
22. Contraindication to anticoagulation
23. Contraindication to isoproterenol
24. Presence of intramural thrombus, tumor or other abnormality that precludes catheter introduction or manipulation
25. Women who are pregnant and/or breast feeding
26. Presence of a condition that precludes vascular access.
27. Patients presenting contraindications for study catheter(s), as indicated in the respective Instructions For Use
28. Enrollment in an investigational study evaluating another device, biologic, or drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Congxin Huang, Principal Investigator — Renmin Hospital of Wuhan University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Sponsor website — https://www.biosensewebster.com/WorldWide/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 201 patients from 12 sites in China were screened and 200 patients were enrolled into the study.
Pre-assignment Details: This was a prospective, multicenter, non-randomized clinical study. Patients were enrolled to receive THERMOCOOL® SMARTTOUCHTM catheter if signed informed consent forms and satisfied the study inclusion and exclusion criteria.
Groups:
- THERMOCOOL® SMARTTOUCH™ Family of Catheters: Pulmonary vein isolation by radiofrequency ablation treatment with the THERMOCOOL® SMARTTOUCH™ contact force sensing catheters (study device)
Period: Overall Study
Arm/Group | THERMOCOOL® SMARTTOUCH™ Family of Catheters
Started (Patients who signed informed consent forms) | 200
Safety Population (All enrolled subjects who underwent insertion of the study catheter) | 200
Intent to Treat (ITT) Population (All enrolled subjects who met the inclusion/exclusion criteria and signed informed consent form) | 193
Per-Protocol Population (ITT subjects with 12 month primary efficacy data and insertion of the study catheter and ablation) | 166
Completed | 185
Not Completed | 15
Not completed — Withdrawal by Subject | 3
Not completed — Death | 1
Not completed — Lost to Follow-up | 11

BASELINE CHARACTERISTICS:
Population: All enrolled subjects
Arm/Group | THERMOCOOL® SMARTTOUCH™ Family of Catheters
Number analyzed (Participants) | 200
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: All enrolled subjects
  Years | 61.2 (9.25)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All enrolled subjects
  Participants
    Female | 75
    Male | 125
Race/Ethnicity, Customized [Number; unit: Participants] — Race/Ethnicity categories related to Chinese are used since the study was conducted in China Population: All enrolled subjects
  Participants
    Han Nationality | 198
    Others: Hui Nationality | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Freedom From Documented Symptomatic Atrial Fibrillation (AF), Atrial Tachycardia (AT), or Atrial Flutter (AFL) Episodes
Description: The primary effectiveness endpoint for this study is freedom from documented symptomatic atrial fibrillation (AF), atrial tachycardia (AT), or atrial flutter (AFL) episodes through 12-month follow-up after the index ablation procedure (includes a three-month blanking period).
Time Frame: 12 Months
Population: Per protocol population: Subjects in the ITT Population who undergone insertion of the study catheter and AF ablation procedure, and had the 12th month primary efficacy endpoint data.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | THERMOCOOL® SMARTTOUCH™ Family of Catheters
Number analyzed (Participants) | 166
Percentage of Participants | 80.7 [73.9 to 86.4]
Statistical Analysis 1: Comparison: THERMOCOOL® SMARTTOUCH™ Family of Catheters; Test type: Other; Proportion of participants = 80.7, 95% CI 2-sided [73.9 to 86.4]; 95% confidence interval is based on Clopper-Pearson confidence interval

2. Secondary Outcome: Percentage of Patients Where Acute Success Was Achieved
Description: Confirmation of entrance block in all pulmonary veins (PVs) with an isoproterenol intravenous challenge 0.5h post procedure. Exit Block is optional for this study.
Time Frame: 0.5 hours
Population: Safety Population, i.e., all enrolled subjects who undergone insertion of the study catheter during the procedure
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | THERMOCOOL® SMARTTOUCH™ Family of Catheters
Number analyzed (Participants) | 200
Percentage of participants | 99.5 [97.2 to 100.0]
Statistical Analysis 1: Comparison: THERMOCOOL® SMARTTOUCH™ Family of Catheters; Test type: Other; Proportion of participants = 99.5, 95% CI 2-sided [97.2 to 100.0]; 95% confidence interval is based on Clopper-Pearson confidence interval

3. Secondary Outcome: Average Contact Force Per Pulmonary Vein Ablation Procedure
Description: Contact force (CF) is the force (g) between the device tip and endocardial wall. Two subjects didn't have CF data
Time Frame: 1 day during procedure
Population: Safety population with contact force data available
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | THERMOCOOL® SMARTTOUCH™ Family of Catheters
Number analyzed (Participants) | 198
Grams | 12.9 (3.79)

4. Secondary Outcome: Percent of Subjects With Pulmonary Vein Reconnection for the Index Procedure
Description: Percentage of subjects with PV reconnection after the first ablation
Time Frame: 1 day during procedure
Population: Safety population with pulmonary vein reconnection data available
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | THERMOCOOL® SMARTTOUCH™ Family of Catheters
Number analyzed (Participants) | 199
Percentage of participants | 7.5 [4.3 to 12.1]

5. Secondary Outcome: Procedure Time, Ablation Time and Fluoroscopy Time
Description: Procedure Time, Ablation Time and Fluoroscopy Time in minutes
Time Frame: 1 day during procedure
Population: Safety population
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | THERMOCOOL® SMARTTOUCH™ Family of Catheters
Number analyzed (Participants) | 200
Minutes
  Duration of Procedure (min) | 144.5 (41.28)
  Duration of Ablation (min) | 63.5 (36.15)
  Total Duration of Fluoroscopy (min) | 15.6 (10.02)

ADVERSE EVENTS:
Time Frame: 12 months after ablation procedure
Arm/Group | THERMOCOOL® SMARTTOUCH™ Family of Catheters
All-Cause Mortality (participants affected / at risk) | 1/200
Serious Adverse Events (participants affected / at risk) | 26/200
Other Adverse Events (participants affected / at risk) | 28/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | THERMOCOOL® SMARTTOUCH™ Family of Catheters (N=200)
Pericardial effusion (Cardiac disorders) | 3 (3)
Pneumonia (Infections and infestations) | 3 (4)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Arteriovenous fistula (Vascular disorders) | 2 (2)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Coronary heart disease (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1)
Syncope (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Mixed connective tissue disease (Musculoskeletal and connective tissue disorders) | 1 (1)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Ischaemia (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1)
Gas poisoning (Injury, poisoning and procedural complications) | 1 (1)
Arteriogram coronary (Investigations) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | THERMOCOOL® SMARTTOUCH™ Family of Catheters (N=200)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 1 (1)
Chest discomfort (General disorders) | 3 (3)
Chest pain (General disorders) | 1 (1)
Ecchymosis (Vascular disorders) | 3 (3)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Haematoma (Vascular disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (6)
Neutrophil count increased (Investigations) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (2)
Pyrexia (General disorders) | 6 (6)
Vessel puncture site haematoma (Vascular disorders) | 3 (3)
Vessel puncture site haemorrhage (Vascular disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4)
Wound secretion (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator (PI)/Institution and the Sponsor (or its agents) that restricts the PI's rights to discuss, present or publish trial results after the trial is completed. Please contact Biosense Webster, Inc. for additional information.

DOCUMENTS (2):
  • Study Protocol (2016-01-07): https://cdn.clinicaltrials.gov/large-docs/25/NCT02485925/Prot_000.pdf
  • Statistical Analysis Plan (2016-05-19): https://cdn.clinicaltrials.gov/large-docs/25/NCT02485925/SAP_001.pdf